CLINICAL TRIAL: NCT02805062
Title: Manometry vs Clinical Assessment in the Detection of Trapped Lung in Patients With Suspected Pleural Malignancy
Acronym: MASCOT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Rocket Medical plc (Other)
Responsible Party: Sponsor
Other Study IDs: GN16ON124
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Pleural Effusion, Malignant
Keywords: Trapped Lung
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pleural Effusion: Malignant pleural effusion patients requiring investigation with thoracoscopy.
  Interventions: Procedure: Digital Pleural Manometry; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Digital Pleural Manometry — Measurement of intra-pleural pressure and the removal of pleural fluid.
Procedure: Magnetic Resonance Imaging — Subject lies a long tunnel shaped scanner and images are recorded.
  Other Names: MRI

SUMMARY:
Malignant pleural effusion is a common clinical problem with median survival of approximately 6 months thus efficient management of Malignant pleural effusion is important. In patients with a Trapped Lung, pleurodesis will be unsuccessful and an indwelling pleural catheter should be inserted instead. Accurate detection of Trapped Lung prior to insertion would avoid futile attempts at talc pleurodesis, re-intervention following failed pleurodesis and allow adequate time to plan for an indwelling pleural catheter insertion.Pleural manometry allows direct and objective measurement of intra-pleural pressure during pleural fluid aspiration.The primary aim of this study is to determine whether the addition of digital pleural manometry to clinical judgment, prior to and during local anaesthetic thoracoscopy, results in a clinically meaningful improvement in Trapped Lung detection.

DETAILED DESCRIPTION:
Malignant pleural effusion is a common clinical problem with median survival of approximately 6 months. Efficient management of Malignant pleural effusion is therefore a major priority for patients, for whom failed procedures and the need for repeat hospital admissions limits their time at home with family and friends.

The management of Malignant pleural effusion involves either complete pleural fluid drainage followed by some form of pleurodesis or insertion of an indwelling pleural catheter. Apposition of the parietal and visceral pleural surfaces is a pre-requisite for successful pleurodesis. In patients with a non-expansile, or Trapped Lung, pleurodesis will be unsuccessful and an indwelling pleural catheter should be inserted instead. Accurate detection of Trapped Lung prior to insertion would avoid futile attempts at talc pleurodesis, re-intervention following failed pleurodesis and allow adequate time to plan for an indwelling pleural catheter insertion, including training of the patient's District Nurses. Clinical judgment is currently used to detect Trapped Lung. This involves review of available imaging and direct visualisation of the surface of the lung during local anaesthetic thoracoscopy. Unfortunately, recent data suggest this is frequently inaccurate, with 30% and 13% of cases of Trapped Lung correctly identified in recent local and national audit data respectively.

Pleural manometry allows direct and objective measurement of intra-pleural pressure during pleural fluid aspiration. Pleural pressure measurements can also be used to compute Pleural Elastance, defined as change in pleural pressure divided by change in pleural volume. Previous studies have shown that a rapid and sustained drop in intra-pleural pressure during fluid aspiration can predict Trapped Lung but these data have not been prospectively compared with current clinical practice.

The primary aim of this study is to determine whether the addition of digital pleural manometry to clinical judgment, prior to and during local anaesthetic thoracoscopy, results in a clinically meaningful improvement in Trapped Lung detection. Digital pleural manometry will be recorded using a Conformité Européene marked (CE-marked) device used within its existing clinical indication (developed in conjunction with our commercial partner Rocket Medical plc).

65 Subjects will have a single study visit, which will coincide with their planned clinical admission for local anaesthetic thoracoscopy. Subjects will exit the study after a follow-up clinic visit 3 months after the date of local anaesthetic thoracoscopy. A study-specific volumetric Magnetic Resonance Imaging scan of the pleural cavity will be performed as per pre-defined imaging protocols.

The study will be performed at a single centre: Queen Elizabeth University Hospital, Glasgow.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* Suspected pleural malignancy requiring investigation by local anaesthetic thoracoscopy

Exclusion Criteria:

* Any contra-indication to local anaesthetic thoracoscopy
* Predicted pleural aspiration volume < 1 litre, as defined by a maximum pleural fluid depth of < 4 cm on thoracic ultrasound pre-aspiration
* Known contra-indication to MRI
* Previous attempt at talc pleurodesis
* Pregnancy
* • Renal impairment (eGFR ≤ 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pleural effusion requiring further investigation with thoracoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pleural Elastance | Single visit per subject
  Pleural elastance (change in pleural pressure divided by change in pleural volume), where trapped lung will be predicted by pleural elastance ≥ 14.5 cm pleural pressure.
Clinical judgement | Single visit per subject
  The clinical judgment of the Thoracoscopist as to the presence or absence of Trapped Lung
Trapped Lung | Single visit per subject
  Occurrence of trapped lung, defined as incomplete lung re-expansion on the pre-discharge chest radiograph after local anaesthetic thoracoscopy

SECONDARY OUTCOMES:
PEL-VOUT Agreement | Single visit per subject
  level of agreement between Indirect Pleural Elastance (PEL) computed using pleural fluid output (VOUT) and Direct PEL, computing using directly measured pleural cavity volume by MRI.

IPD SHARING:
Plan to Share IPD: No
Published results will not personally identify study subjects.